CLINICAL TRIAL: NCT05103891
Title: A Randomized, Single-center, Open-label, Single Dose, Two-period, Crossover Study to Investigate the Relative Bioavailability of Binimetinib 3 x15 mg and 45 mg Tablets in Healthy Participants
Brief Title: Relative Bioavailability of Binimetinib 3 x 15 mg and 45 mg Formulations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: W00074CI101_1PF73
Record Dates: First submitted 2021-09-29; First posted 2021-11-02 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Melanoma; BRAF V600 Mutation; Unresectable Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binimetinib 15 mg / Binimetinib 45 mg (Experimental): 2 periods
  Interventions: Drug: Binimetinib Oral Tablet
- Binimetinib 45 mg / Binimetinib 15 mg (Experimental): 2 periods
  Interventions: Drug: Binimetinib Oral Tablet

INTERVENTIONS:
Drug: Binimetinib Oral Tablet — two-period, crossover study

SUMMARY:
The current commercially available MEKTOVI® (binimetinib) 15 mg tablets are provided as immediate release film-coated tablets for oral administration. For the treatment of adult patients with unresectable or metastatic melanoma with BRAF V600 mutation, the recommended dosing regimen is 45 mg twice daily (bis in die, BID). No food effect with the commercial formulation of 15 mg was demonstrated.

In order to reduce the patient's burden, a new strength tablet containing 45 mg of binimetinib as active ingredient is being developed. As a result, the number of tablets to be taken by the patients will be reduced from 6 tablets (6 x 15 mg) to 2 tablets (2 x 45 mg) per day. The evaluation of the relative bioavailability of the 45 mg tablet in comparison to three 15 mg tablets intake is therefore required.

DETAILED DESCRIPTION:
The R formulation is the currently commercially available tablet containing 15 mg of binimetinib as active substance, administered as three tablets for a total of 45 mg binimetinib. The T formulation is the tablet containing 45 mg of binimetinib as active substance in one tablet. Participants will be randomized to one of 2 treatment sequences (RT or TR) containing 2 treatment periods, with at least a 7-day washout between each dose.

The study will consist of a screening period between 21 and 2 days before the first study treatment administration on Period (P) 1 Day (D) 1, 2 treatment periods of 5 days each, and a washout of at least 7 days between P1D1 and P2D1.

Study treatments are given by the oral route in fasted condition. The end-of-study (EOS) visit will be performed 30 (± 3) days after the last study treatment administration or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participant.
2. Female participants must be postmenopausal or sterilized.
3. Body mass index (BMI) of ≥ 18.5 to < 30 kg/m2, with body weight ≥ 50 kg and < 100 kg.
4. Vital signs within the following ranges or if out of normal ranges, considered as not clinically significant by the Investigator.
5. Participants must have safety laboratory values within the normal ranges or if out of normal ranges considered as not clinically significant by the Investigator.

Exclusion Criteria:

1. Pregnant or currently breastfeeding women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
2. A past medical history of clinically significant ECG abnormalities or a family history (grandparents, parents, and siblings) of prolonged QT interval syndrome.
3. Impaired cardiovascular function.
4. History of fainting spells or orthostatic hypotension episodes.
5. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the participant in case of participation in the study.
6. History of autonomic dysfunction or Gilbert syndrome.
7. History or current evidence of Central serous retinopathy (CSR), Retinal vein occlusion (RVO) or ophthalmopathy as assessed by ophthalmologic examination at baseline that would be considered a risk factor for CSR/RVO [e.g., optic disc cupping, visual field defects, intraocular pressure (IOP) > 21 mmHg].
8. Neuromuscular disorders that were associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
9. Smoker or use of tobacco products or products containing nicotine in the last 4 weeks prior to first dosing of study treatment.
10. Malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma of the skin (adequate wound healing is required prior to study entry).
    2. Primary malignancy which had been completely resected and was in complete remission for ≥ 5 years.
11. History of retinal degenerative disease.
12. Any vaccination within 4 weeks prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2021-11-29 (Estimated); Study Completion 2021-11-29 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time of administration to last observed plasma concentration (AUClast) | Through study completion, an average of 2 months
AUC from time of administration to infinity (AUCinf) | Through study completion, an average of 2 months
Maximum observed plasma concentration (Cmax) | Through study completion, an average of 2 months
Time to reach Cmax (Tmax) | Through study completion, an average of 2 months
AUC Test(T) / Reference (R) ratios | Through study completion, an average of 2 months

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Through study completion, an average of 2 months
  Incidence, nature and severity
Treatment-emergent serious adverse events (treatment-emergent SAEs) | Through study completion, an average of 2 months
  Incidence, nature and severity
Electrocardiograms | Through study completion, an average of 2 months
  heart rate (HR), PR interval, QRS duration, QRS axis, QT interval, QTcF
Clinical laboratory parameters | Through study completion, an average of 2 months
  Erythrocytes (red blood cells, RBCs), hematocrit, hemoglobin, platelets; leukocyte count with differential: basophils, eosinophils, lymphocytes, monocytes, neutrophils / absolute neutrophil count; RBC indices: mean corpuscular hemoglobin, mean corpuscular volume, reticulocytes/erythrocytes, ALT, albumin, ALP, AST, bicarbonate, bilirubin (total and indirect), urea, calcium, chloride, CK, creatinine, amylase, lipase, total cholesterol, glucose, lactate dehydrogenase, magnesium, potassium, sodium, total protein, uric acid, blood pregnancy test (hCG), coagulation (aPTT or PT)
Vital signs | Through study completion, an average of 2 months
  Supine and standing systolic BP, diastolic BP and PR, body temperature
Opthalmologic examinations | At the screening and at the end of study
  Best corrected visual acuity for distance testing, optical coherence tomography and/or fluorescein angiography, slit lamp examination, IOP and dilated fundoscopy with attention to retinal abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Marina Klein, MD, Principal Investigator — Biotrial
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: No